CLINICAL TRIAL: NCT00162643
Title: Boosted PI VS. NNRTI Based Therapy as Initial Treatment for HIV-1 Infected Patients With Advanced Disease
Brief Title: PI Vs. NNRTI Based Therapy for HIV Advanced Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Collaborators: National Council of Science and Technology, Mexico (Other); Instituto Mexicano del Seguro Social (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SALUD-2003-C01-123
Record Dates: First submitted 2005-09-07; First posted 2005-09-13 (Estimated); Last update posted 2006-09-14 (Estimated); Status verified 2006-09

CONDITIONS: Acquired Immunodeficiency Syndrome
Keywords: Acquired Immunodeficiency Syndrome; Antiretroviral Therapy, Highly Active; Protease Inhibitors; Reverse Transcriptase Inhibitors
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Ritonavir; Zidovudine; Lamivudine; efavirenz

INTERVENTIONS:
Drug: zidovudine+lamivudine+lopinavir/ritonavir
Drug: zidovudine + lamivudine + efavirenz

SUMMARY:
Ritonavir boosted protease inhibitor based therapy will have equivalent antiviral efficacy over 48 weeks compared to NNRTI based therapy in patients who are antiretroviral therapy naïve and initiate therapy with CD4 counts ≤ 200/mm3.

DETAILED DESCRIPTION:
Current guidelines for initial therapy in HIV infection recommend 2 NRTIs plus either a ritonavir boosted protease inhibitor or a non-nucleoside reverse transcriptase inhibitor (NNRTI). Recent data suggests that the rate of response to PI based therapy may be slightly compromised if the baseline CD4 count is ≤ 200/mm3 and the plasma HIV-1-RNA ≥ 100,000 copies/mL. This may not be equally apparent if ritonavir boosted protease inhibitors are used. The effect of baseline CD4 count and HIV-1-RNA levels on the antiviral efficacy of NNRTI based regimens has been less well characterized. A significant number of patients currently initiate therapy at late stages of progression, typically with baseline CD4 count is ≤ 200/mm3. In Mexico approximately 60% of patients who initiate therapy are within this range of CD4 cell counts. Currently, the two combinations recommended as preferred are with two NRTIs and either Efavirenz or Lopinavir/ritonavir, while other combinations of PIs and ritonavir are considered alternative.

Comparison: The efficacy of ritonavir boosted protease inhibitor based therapy versus NNRTI based therapy in patients who are antiretroviral therapy naïve and initiate therapy with a CD4 count ≤ 200/mm3.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected individuals
* Men or women at least 18 years old
* CD4+ T cells ≤200/ml
* Antiretroviral naive

Exclusion Criteria:

* Suspected or documented active, untreated HIV 1 related opportunistic infection (OI) or other condition requiring acute therapy (e.g., hepatitis C virus infection)
* Platelet count < 75,000 cells/mm3.
* Hemoglobin < 9 g/dL .
* AST and/or ALT greater than 5 times the upper limit of normal
* Documented or suspected active tuberculosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2004-12; Study Completion 2007-12

PRIMARY OUTCOMES:
Percentage of patients who reach HIV-1-RNA ≤ 50 copies/mL at 48 weeks

SECONDARY OUTCOMES:
plasma Viral Load change from baseline
Clinical symptoms
CD4 counts
Safety
Tolerability
Discontinuations

CONTACTS AND LOCATIONS:
Overall Officials: Juan G Sierra-Madero, MD, Study Chair — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Locations (5):
- Mexico (5):
  - Hospital de Especialidades Centro Medico Nacional siglo XXI, Mexico City, D.F.
  - Hospital General Regional de Leon, León, Guanajuato
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, Mexico City, Mexico City
  - Hospital General Regional #53, Los Reyes Acaquilpan, State of Mexico
  - Hospital General Regional #72, Tlalnepantla, State of Mexico

REFERENCES:
- [Derived] Lima VD, Sierra-Madero J, Wu Z, Singer J, Wood E, Hull MW, Richard Harrigan P, Montaner JS. Comparing the efficacy of efavirenz and boosted lopinavir using viremia copy-years. J Int AIDS Soc. 2014 May 6;17(1):18617. doi: 10.7448/IAS.17.1.18617. eCollection 2014. PMID 24805184